CLINICAL TRIAL: NCT05449691
Title: BIOSYM - A Feasibility Randomised Controlled Trial Comparing Biological Matrices With Synthetic Meshes in Women Undergoing One Stage Implant Based Breast Reconstruction
Brief Title: Biological Matrices Versus Synthetic Meshes
Acronym: BIOSYM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Amit Goyal, Chief Investigator, University Hospitals of Derby and Burton NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 315581
Record Dates: First submitted 2022-07-04; First posted 2022-07-08 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: breast reconstruction; mesh; acellular dermal matrix; synthetic mesh; breast cancer; patient reported outcome
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biological Matrix (Active Comparator): Participants will undergo immediate breast reconstruction using biological matrix and implant
  Interventions: Procedure: One-stage immediate breast reconstruction
- Synthetic Mesh (Experimental): Participants will undergo immediate breast reconstruction using synthetic mesh and implant
  Interventions: Procedure: One-stage immediate breast reconstruction

INTERVENTIONS:
Procedure: One-stage immediate breast reconstruction — One-stage mesh assisted implant breast reconstruction

SUMMARY:
In this feasibility study, 60 women undergoing reconstruction will be randomly allocated to receive biological or synthetic mesh and followed for 6 months. The findings will tell us if patients and surgeons are comfortable with not being able to choose which mesh is used for the operation. In the larger surgical study, the investigators plan to measure patients' satisfaction with the reconstruction, patients' quality of life, complications from the operation and costs over 5 years.

DETAILED DESCRIPTION:
Immediate breast reconstruction in women undergoing removal of the whole breast for cancer or risk reduction is most commonly done using breast implants. Surgeons often use a sheet of mesh to cover the implant as standard treatment. It acts like an internal bra and supports the implant and re-creates a natural looking breast.

Natural(biological) or man-made (synthetic) meshes are used routinely in the NHS. Biological ones are made from animal tissue (pig, cow) that have been made safe to use in people and are costly. Synthetic meshes are made from net-like fabric and cost less. The choice about which mesh to use depends on surgeons' personal experience and how much money the hospital has for these operations. The two meshes may have different acceptability issues for patients because of their personal values, religious beliefs, ethnic background or views on animal welfare.

A large UK review of breast reconstruction with implants gathered information up to 3 months after surgery on the use and outcomes of the two meshes. This suggests that both may be equally safe in the short-term. However, this information can be improved by comparing the meshes side-by-side and looking at how safe they are long-term. This is important as some side-effects only appear later after surgery. Clinicians do not know how outcomes impact on patients' health and well-being.

The best proof would come from a randomised surgical study, where a computer allocates patients to receive either the biological or synthetic mesh. Investigators will measure how patients feel, how their health is, and record if they have any side-effects from the reconstructive surgery. This type of study would tell us how good each mesh is and if they are safe long-term.

Before starting such a study, investigators will run a smaller one that will help us understand if patients and surgeons would be comfortable taking part.

ELIGIBILITY:
Inclusion Criteria:

Female age ≥ 18 Women undergoing mastectomy and immediate one-stage mesh assisted implant breast reconstruction as standard treatment

Exclusion Criteria:

Revision reconstruction surgery Delayed reconstruction surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinician acceptance | 2 years
  Proportion of eligible women offered the trial
Patient acceptance | 2 years
  Proportion of women offered the trial who participate in the trial
Recruitment rate | 2 years
  Number of patient recruited per year per site
Compliance with allocated intervention | 2 years
  Number of patients not complying with randomisation allocation

CONTACTS AND LOCATIONS:
Overall Officials: Amit Goyal, MS, MD, FRCS, Study Chair — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (5):
- United Kingdom (5):
  - University Hospitals of Derby and Burton NHS Foundation Trust, Derby
  - Wycombe Hospital, High Wycombe
  - Castle Hill Hospital, Hull
  - University Hospitals of Leicester NHS Trust, Leicester
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2025-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT05449691/Prot_000.pdf